CLINICAL TRIAL: NCT04381377
Title: A Multi-centre, Adaptive, Randomized, Double-blind, Placebo-controlled Comparative Clinical Study of the Safety and Efficacy of Polyoxidonium®, Lyophilizate for Solution for Injections and Topical Application, 6 mg (NPO Petrovax Pharm LLC, Russia) in Patients With Coronavirus Disease (COVID-19).
Brief Title: Efficacy and Safety of Polyoxidonium® in Hospitalized Patients With Coronavirus Disease COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NPO Petrovax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PО-COV-III-20
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Infections, Coronavirus
Keywords: COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — azoximer bromide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyoxidonium (Experimental): Polyoxidonium will be administered in the dose of 12 mg (contents of 2 vials) once daily intravenously (IV) for 3 days, then every other day intramuscularly (IM) on days 5-17 (the total treatment course is 10 injections).
  Interventions: Drug: azoximer bromide
- Placebo (Placebo Comparator): Placebo will be administered (contents of 2 vials) once daily intravenously (IV) for 3 days, then every other day intramuscularly (IM) on days 5-17 (the total treatment course is 10 injections).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: azoximer bromide — Investigational medicinal product
  Other Names: Polyoxidonium
  Arms: Polyoxidonium
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the superiority of Polyoxidonium®, lyophilizate for solution for injections and topical application, 6 mg over placebo in hospitalized patients with coronavirus disease (COVID-19). This is a multicentre prospective, randomized, double-blind, placebo-controlled, parallel-group phase IIb\IIIa clinical trial.

DETAILED DESCRIPTION:
This is a multicenter prospective, randomized, double-blind, placebo-controlled, parallel-group phase 3 IIb\IIIa trial to evaluate the efficacy of Polyoxidonium®, lyophilizate for solution for injections and topical application, 6 mg over placebo in hospitalized patients with coronavirus disease (COVID-19). A study will last for 29±3 days (maximum) for each participant and will include: screening (days -1...1); treatment period (17 days in total, days 1...17) with the administration of the investigational product Polyoxidonium/placebo (intravenous injections for 3 days, then intramuscular injections for 14 days), assessment of the clinical status, recording of AEs; follow-up period (days 18...29±3).

Haematology and blood chemistry tests will be performed at day -1 and days 1,3, 8 ±1, 17±1.

Assessment of the clinical status according to the 7-point ordinal scale and according to the National Early Warning Score (NEWS) scale will be done every day during hospitalization from day 1 up to and including day 17 and at the follow-up on day 29±3.

The safety and tolerability will be evaluated throughout the study (from signing the Informed Consent Form to the study completion visit).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients from 18 to 85 years of age.
2. The patient (or his/her legal representative, if the patient is not able to sign the form) signed an Informed Consent form for participation in this study before any initiation of any study procedures.
3. The patient can understand all protocol requirements, perform the study procedures, and agree to all limitations specified in the protocol.
4. Confirmed diagnosis of coronavirus disease (COVID-19): laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other commercial or public health assay in any specimen < 14 days prior to randomization.
5. Illness (coronavirus disease COVID-19) of any duration, and at least one of the following:

   * Radiographic/tomographic chest infiltrates by imaging (chest x-ray, CT scan, etc.), OR
   * Evidence of rales/crackles on clinical exam AND SpO2 ≤ 94% on room air, OR
   * Indications for mechanical ventilation and/or supplemental oxygen.
6. Agrees to use adequate contraception methods (the methods with at least 90% efficacy include non-hormonal intrauterine devices; condom with intravaginal spermicide; cervical caps

Exclusion Criteria:

1. History of clinically significant allergic reactions.
2. Hypersensitivity and/or intolerability to any ingredient of the investigational product or placebo.
3. Anticipated transfer to another hospital which is not a study centre within the next 72 hours.
4. Acute or chronic renal failure.
5. History of HIV infection, tuberculosis.
6. Conditions associated with primary immunodeficiency.
7. Concomitant use of cytostatic medications to treat a concomitant disease.
8. Systemic connective tissue diseases.
9. Need for the prohibited medications.
10. Administration of medications that are prohibited or unauthorized by the protocol within 2 weeks before the expected randomization date.
11. History of alcohol or drug dependence.
12. History of malignant tumours of any location with remission for less than 2 years.
13. History of psychic (including depressive) disorders, physical and other factors that do not allow for adequate self-assessment of one's behaviour and for compliance with the protocol requirements, including history of psychiatric disorders.
14. Pregnancy or breastfeeding.
15. Intravenous injections and/or sampling of the required amount of blood is not possible.
16. Positive pregnancy test (in patients with childbearing potential).
17. Participation in any clinical study within 3 months before enrolment in this study.
18. History of any condition that the study doctor considers significant enough to prevent enrolment of this patient.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Clinical status of the patient (according to 7-point ordinal scale) | Day 15
  The primary efficacy outcome will be defined based on the blinded analysis of data of the first 100 patients in the 1st part of the study. There is uncertainty about the clinical course and potential different trajectories according to baseline disease severity, so the day of the primary endpoint may be modified based on a blinded evaluation of the primary efficacy outcome in various days.

SECONDARY OUTCOMES:
Clinical status of the patient (according to 7-point ordinal scale) | Clinical status of the patient and the average change in the ordinal scale from baseline, both on days 3, 5, 8, 11, 29.
  Time to improvement by one category from admission on the ordinal scale. Clinical status of the patient. Average change in the ordinal scale from baseline.
NEWS | Change in NEWS from baseline on days 3, 5, 8, 11, 15, 29.
  The time to discharge or to a NEWS of ≤ 2 and maintained for 24 hours, whichever occurs first.
  Change in NEWS from baseline.
Oxygenation | Oxygenation free days in the first 28 days (to day 29). Incidence and duration of new oxygen use during the study.
  Oxygenation free days. Incidence and duration of new oxygen use.
Mechanical Ventilation | Ventilator free days in the first 28 days (to day 29). Incidence and duration of new mechanical ventilation use during the trial.
  Ventilator free days. Incidence and duration of new mechanical ventilation use.
Mortality | 28-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Rossi, Professor, Principal Investigator — University of Montpellier (Faculté de Médecine) and Institute Sainte Catherine
Locations (14):
- Russia (12):
  - Regional state budgetary institution of public health "City hospital No. 5 of Barnaul", Barnaul
  - Central Research Institute of Epidemiology of Rospotrebnadzor, Moscow
  - The state healthcare institution of the city of Moscow "City Clinical Hospital No. 15 named after OM Filatov" in "Moscow City Department of Health", Moscow
  - Moscow State Budgetary Healthcare Institution "Infectious Clinical Hospital No. 1 of the Moscow Department of Healthcare", Moscow
  - Moscow State Budgetary Healthcare Institution "City Clinical Hospital No. 24 of the Moscow Department of Healthcare", Moscow
  - State budgetary institution "Research Institute of Emergency Care named after N.V. Sklifosovsky in Department of Health of the city of Moscow", Moscow
  - Moscow State Budgetary Healthcare Institution "City Clinical Hospital No. 40 of the Moscow Department of Healthcare", Moscow
  - State budgetary institution of health care of the Nizhny Novgorod region "Infectious clinical hospital No. 2 of Nizhny Novgorod", Nizhny Novgorod
  - Federal State Budgetary Educational Institution of Higher Education "Orenburg State Medical University" of the Ministry of Health of the Russian Federation, Orenburg
  - Federal State Budgetary Educational Institution of Higher Education "First St. Petersburg State Medical University named after Academician I.P. Pavlov, Saint Petersburg
  - State budgetary health institution of the Vladimir region "Regional Clinical Hospital", Vladimir
  - Yaroslavl State Medical University of Ministry of Health of the Russian Federation, Yaroslavl
- Slovakia (2):
  - Clinics of Infectious Diseases, University Hospital in Nitra, Nitra
  - Clinics of Infectious Diseases, University Hospital in Trnava, Trnava